CLINICAL TRIAL: NCT02303353
Title: Data Base Project for Acquisition of Cancer Patient Data in Practices and Ambulant Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: SPGO Research Mannheim GmbH (Industry)
Collaborators: AKP Freiburg GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: REGONKO-01
Record Dates: First submitted 2014-11-03; First posted 2014-11-27 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Carcinoma
Keywords: Breast cancer; Ovarian cancer; Lung cancer; Colon cancer; Gastric cancer; Pancreatic cancer; Rectum cancer; Plasmacytoma
MeSH Terms: conditions — Carcinoma; Breast Neoplasms; Ovarian Neoplasms; Lung Neoplasms; Colonic Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Rectal Neoplasms; Plasmacytoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cancer patients: Patients suffering from a carcinoma (either breast, ovarian, lung, colon, stomach, pancreas, rectum or plasmacytoma)

SUMMARY:
The purpose of this registry is to evaluate the situation regarding ambulant therapy of cancer patients in different practices in Germany. It should provide insight into the implementation of schemes for cancer therapy predefined in the guidelines, the treatment of diverse adverse reactions and the counter measures taken. Thereby, potential differences in treatment and with that differences in quality amongst individual practices might be identified. The medium to long term aim is to contribute to positively influence the quality of medical care of cancer patients in Germany.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Tumor disease (carcinoma of either breast, ovary, lung, colon, stomach, pancreas, rectum or plasmacytoma)
* Written informed consent

Exclusion Criteria: none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from carcinoma which are treated in practices (ambulant therapy)
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2013-10; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Anti-cancer treatments (Course of the disease and type of applied anti-cancer therapies. Assessment of guidelines' implementation) | From date of ICF until date of cure/death/ICF withdrawal, up to 60 months
  Course of the disease and type of applied anti-cancer therapies. Assessment of guidelines' implementation

SECONDARY OUTCOMES:
Adverse reactions and their treatment (Number and type of adverse reactions and applied counter measures / therapies) | From date of ICF until date of cure/death/ICF withdrawal, up to 60 months
  Number and type of adverse reactions and applied counter measures / therapies

CONTACTS AND LOCATIONS:
Locations (1):
- Practice, Mannheim, Germany